CLINICAL TRIAL: NCT03714737
Title: Immunogenicity and Safety of Bivalent Meningococcal Serogroups A and C Tetanus Toxoid Conjugate Vaccine in Chinese Healthy Children Aged 3 Months to 5 Years.: A Randomized, Blinded, Positive Controlled Phase III Clinical Trial
Brief Title: Immunogenicity and Safety of Bivalent Meningococcal Serogroups A and C Tetanus Toxoid Conjugate Vaccine in Chinese
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JSVCT028
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Experimental 1 (Experimental): Experimental vaccine of 0.5ml in 300 children aged 2-5 years at day 0.
  Interventions: Biological: experimental vaccine
- Positive control 1 (Active Comparator): Positive control vaccine 1 of 0.5ml in 300 children aged 2-5 years at day 0.
  Interventions: Biological: Positive control vaccine 1
- Experimental 2 (Experimental): Experimental vaccine of 0.5ml in 150 children aged 12-23 months at day 0 and 28.
  Interventions: Biological: experimental vaccine
- Experimental 3 (Experimental): Positive control vaccine 2 of 0.5ml in 150 children aged 12-23 months at day 0.
  Interventions: Biological: experimental vaccine
- Positive control 2 (Active Comparator): Positive control vaccine 2 of 0.5ml in 150 children aged 12-23 months at day 0 and 28.
  Interventions: Biological: Positive control vaccine 2
- Experimental 4 (Experimental): Experimental vaccine of 0.5ml in 150 children aged 2-5 years at day 0 and 28, and boost at 18 months.
  Interventions: Biological: experimental vaccine
- Positive Control 3 (Active Comparator): Positive control vaccine 2 of 0.5ml in 150 children aged 6-11 months at day 0 and 28.
  Interventions: Biological: Positive control vaccine 2
- Experimental 5 (Experimental): Experimental vaccine of 0.5ml in 300 children aged 3-5 months at day 0, 28, 56, and boost at 18 months.
  Interventions: Biological: experimental vaccine
- Positive Control 4 (Active Comparator): Positive control vaccine 1 of 0.5ml in 300 children aged 3-5 months day 0, 28, 56.
  Interventions: Biological: Positive control vaccine 1

INTERVENTIONS:
Biological: experimental vaccine — bivalent meningococcal serogroups A and C tetanus toxoid conjugate vaccine(OLYMVAX Biological Co., LTD)
  Arms: Experimental 1; Experimental 2; Experimental 3; Experimental 4; Experimental 5
Biological: Positive control vaccine 1 — bivalent meningococcal serogroups A and C tetanus toxoid conjugate vaccine(WALVAX Biological Co., LTD)
  Arms: Positive Control 4; Positive control 1
Biological: Positive control vaccine 2 — bivalent meningococcal serogroups A and C tetanus toxoid conjugate vaccine(Royal (Wuxi) Biological Co., LTD)
  Arms: Positive Control 3; Positive control 2

SUMMARY:
Invasive meningococcal disease and meningococcal meningitis caused by Neisseria meningitidis have their highest incidence in children, with a second peak in adolescents and young adults. The most important disease-causing serogroups are meningococcal serogroups A (MenA) and MenC in Asia, such as China. The specific vaccine use in each country depends on the predominant serogroups, cost, and availability. conjugate vaccines are preferred to polysaccharide vaccines due to their impact on decreasing nasopharyngeal carriage of N. meningitidis and their overall increased immunogenicity in children. This clinical trial is planning to evaluate the immunogenicity and safety of bivalent meningococcal serogroups A and C tetanus toxoid conjugate vaccine in Chinese healthy children aged 3 months to 5 years.

DETAILED DESCRIPTION:
Invasive meningococcal disease and meningococcal meningitis caused by Neisseria meningitidis have their highest incidence in children, with a second peak in adolescents and young adults. The most important disease-causing serogroups are meningococcal serogroups A (MenA), MenB, MenC, MenW and MenY. Their prevalence varies geographically, MenA and MenC being more prominent in Asia. Neisseria meningitidis is one of the leading causes of bacterial meningitis globally. The annual number of cases related to invasive meningococcal disease (IMD) is estimated to be at least 1.2 million with 135 000 deaths.1 To combat IMD, an increasing number of countries have included vaccines against N. meningitidis in their routine immunization programs. The specific vaccine use in each country depends on the predominant serogroups, cost, and availability. Polysaccharide vaccines were used in high risk people in Saudi Arabia and Syria and in routine immunization in China and Egypt. In general, conjugate vaccines are preferred to polysaccharide vaccines due to their impact on decreasing nasopharyngeal carriage of N. meningitidis and their overall increased immunogenicity in children. This clinical trial is planning to evaluate the immunogenicity and safety of bivalent meningococcal serogroups A and C tetanus toxoid conjugate vaccine in Chinese healthy children aged 3 months to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 months old group
* Healthy infants aged 3-5months old as established by medical history and clinical examination
* Subjects who was never administered meningococcal vaccine.
* The subjects' guardians are able to understand and sign the informed consent
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature ≤37.0°C on axillary setting 6-23 months old group
* Healthy infants aged 6-23 months old as established by medical history and clinical examination
* Subjects who was never administered meningococcal conjugate vaccine, or administered meningococcal polysaccharide vaccine over 3 months.
* The subjects' guardians are able to understand and sign the informed consent
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature ≤37.0°C on axillary setting 2-5 years old group
* Healthy infants aged 2-5 years as established by medical history and clinical examination
* Subjects who was never administered meningococcal conjugate vaccine, or administered meningococcal polysaccharide vaccine over 12 months.
* The subjects' guardians are able to understand and sign the informed consent
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature ≤37.0°C on axillary setting

Exclusion Criteria:

* Subjects who has a medical history of invasive meningococcal disease and meningococcal meningitis.
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Severe malnutrition or dysgenopathy
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with injections or blood draws
* Any acute infections in last 3 days
* Any prior administration of immunodepressant or corticosteroids in last 14 days
* Any prior administration of attenuated live vaccine in last 14 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Had fever before vaccination, Subjects with temperature >37.0°C on axillary setting
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Exclusion Criteria for the second and third dose:

If Subjects who have one condition as followed, prohibiting to continue the vaccination, and they will be continue observed in the opinion of the investigator. All participants with adverse events as followed, must be settled in follow-up to the end of events.

* Any serious adverse events caused by vaccination.
* Any confirmed or suspected autoimmune diseases or immune deficiency disorders, including human immunodeficiency virus (HIV) infection
* Have acute or new chronic disease during vaccination
* Other reactions that in the opinion of the investigator ( include: severely serious symptom of pain, swelling, Limitation of motion, continuous high fever, headache and other Systemic or local reactions )

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1950 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
seroconversion rates of antibodies after vaccination | 28 days after vaccination
  seroconversion rates of antibodies against meningococcal serogroups A and C
Proportion of subjects reporting solicited injection-site reactions, solicited systemic reactions | Day 7 post-each dose
  Proportion of subjects reporting solicited injection-site reactions, solicited systemic reactions within 7 days post-each dose

SECONDARY OUTCOMES:
Percentage of rSBA titers ≥1:128 and ≥1:8, and GMT for meningococcal serogroups A and C after vaccination in children aged 2-5 years. | 28 days after vaccination
  Percentage of rSBA titers ≥1:128 and ≥1:8, and GMT for meningococcal serogroups A and C at day 28 post vaccination in children aged 2-5 years.
Percentage of rSBA titers ≥1:128 and ≥1:8, and GMT for meningococcal serogroups A and C after vaccination in children aged 12-23 months. | 28 days after vaccination
  Percentage of rSBA titers ≥1:128 and ≥1:8, and GMT for meningococcal serogroups A and C after vaccination in children aged 12-23 months with two vaccination schedules.
Percentage of rSBA titers ≥1:128 and ≥1:8, and GMT for meningococcal serogroups A and C after vaccination in children aged 6-11 months. | 28 days after vaccination
  Percentage of rSBA titers ≥1:128 and ≥1:8, and GMT for meningococcal serogroups A and C after vaccination in children aged 6-11 months.
Percentage of rSBA titers ≥1:128 and ≥1:8, and GMT for meningococcal serogroups A and C after vaccination in children aged 3-5 months. | 28 days after vaccination
  Percentage of rSBA titers ≥1:128 and ≥1:8, and GMT for meningococcal serogroups A and C after vaccination in children aged 3-5 months.
Proportion of subjects reporting unsolicited adverse events | 28 days after vaccination
  Proportion of subjects reporting unsolicited adverse events
Proportion of subjects with Serious Adverse Events occurring throughout the trial | 28 days after vaccination
  Proportion of subjects with Serious Adverse Events occurring throughout the trial

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu J, Li H, Chu K, Liang Q, Li J, Luo L, Hu Y, Meng F, Zhu F. Immunogenicity and safety of a meningococcal serogroups A and C tetanus toxoid conjugate vaccine (MenAC-TT): two immune schedules in toddles aged 12-23 months in China. Hum Vaccin Immunother. 2019;15(12):2952-2959. doi: 10.1080/21645515.2019.1627816. Epub 2019 Jul 26. PMID 31348731